CLINICAL TRIAL: NCT06022523
Title: Accuracy of Pulse Oximeters With Profound Hypoxia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Consolidated Research, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 21-344376
Record Dates: First submitted 2022-11-30; First posted 2023-09-05 (Actual); Last update posted 2023-09-05 (Actual); Status verified 2023-08

CONDITIONS: Hypoxemia
Keywords: Hypoxia; Pulse oximetry
MeSH Terms: conditions — Hypoxia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Acquisition (Experimental): Subjects will undergo profound hypoxia with stable plateaus.
  Interventions: Diagnostic Test: Data acquisition using DT-400 pulse oximetry system

INTERVENTIONS:
Diagnostic Test: Data acquisition using DT-400 pulse oximetry system — Acquisition of photopleth data during profound hypoxia using a Consolidated Research DT-400 pulse oximetry system.

SUMMARY:
The goal of this clinical trial is the acquisition of photoplethysmography signals during periods of profound hypoxia. The study is designed in accordance with ISO 80601- 2-61,2ed:2017-12 & 2018-02.

ELIGIBILITY:
Inclusion Criteria:

-

Exclusion Criteria:

Pregnancy -

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-11-09 (Actual); Primary Completion 2024-11-09 (Estimated); Study Completion 2024-11-09 (Estimated)

PRIMARY OUTCOMES:
Saturation level measurement | Within 12 months of subject recruitment
  Induction of hypoxia by having subjects breathe mixtures of nitrogen, room air, and carbon dioxide to allow measurement of oxyhemoglobin saturation between 70-100%. Each plateau level of oxyhemoglobin saturation was maintained for at least 30 seconds or until reference pulse oximeters readings were stable

CONTACTS AND LOCATIONS:
Locations (1):
- Consolidated Research, Inc., Cleveland, Ohio, United States